CLINICAL TRIAL: NCT07392437
Title: Prevalence of Diabetes-related Distress Among Patients Living With Type 2 Diabetes in a University Hospital Center and Identification of Its Associated Factors.
Acronym: DIAMIND
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 25-PP-21
Record Dates: First submitted 2026-01-08; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Diabetes Mellitus; Psychological Distress
MeSH Terms: conditions — Diabetes Mellitus | interventions — Surveys and Questionnaires; Restraint, Physical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients (Other)
  Interventions: Behavioral: Questionnaire and Physical Exam

INTERVENTIONS:
Behavioral: Questionnaire and Physical Exam — Patients will be asked to complete questionnaires.

SUMMARY:
Diabetes-related distress is a psychological construct associated with poorer glycaemic control in people living with diabetes. In France, few data are available on this topic and none focus specifically on adults with type 2 diabetes. Diabetes-related distress is not mentioned in the current French national guidelines on the management of type 2 diabetes, whereas international societies such as the ADA and, more recently, the EASD now recommend its regular assessment.

This single-centre observational study conducted in the endocrinology department of Nice University Hospital aims to estimate the prevalence of severe diabetes-related distress in adults with type 2 diabetes receiving usual care, and to identify associated clinical, psychosocial and lifestyle factors. Participants complete validated self-report questionnaires (PAID-20 for diabetes distress, WHOQOL-BREF for quality of life, and a modified Starting The Conversation dietary questionnaire), and clinical data are extracted from electronic medical records. The study does not modify usual medical management and participation consists only in completing the questionnaires and receiving feedback on the results.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age ≥ 18 years).
* Diagnosed with type 2 diabetes according to national (HAS) criteria, whether newly diagnosed or longstanding, with or without chronic complications, and with no restriction regarding HbA1c level. Managed for type 2 diabetes in the endocrinology department of Nice University Hospital (conventional hospitalization, day hospital, or outpatient consultation).
* Able to understand the study information and to complete the self-administered questionnaires.
* Affiliated to the French social security system.
* Has not objected to participation in the study (non-opposition procedure).

Exclusion Criteria:

* Age < 18 years.
* Pregnant woman.
* Any type of diabetes other than type 2 diabetes (e.g. type 1 diabetes, secondary or genetic diabetes).
* Haemochromatosis.
* Cystic fibrosis.
* Current treatment with one of the following hyperglycaemic therapies: oral corticosteroids, immunosuppressive drugs, dopaminergic agonists, interferon-alpha, or protease inhibitors.
* History of partial or total pancreatectomy.
* Ongoing genetic work-up for atypical diabetes.
* Non-French-speaking patient.
* Major neurocognitive disorder or physical/mental disability preventing completion of the questionnaires.
* Adult under legal protection (guardianship or curatorship).
* Refusal or subsequent withdrawal of non-opposition.
* Any later paraclinical result finally revealing a type of diabetes other than type 2 diabetes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Estimated)
Dates: Start 2026-03-02 (Estimated); Primary Completion 2027-01-02 (Estimated); Study Completion 2027-01-02 (Estimated)

PRIMARY OUTCOMES:
Prevalence of severe diabetes-related distress (PAID-20 score ≥ 40) | Baseline (single assessment during usual care visit, within 3 days from inclusion)
  Diabetes-related distress will be assessed using the Problem Areas In Diabetes scale (PAID-20). The PAID-20 includes 20 items scored from 0 to 4; the total raw score (0-80) is multiplied by 1.25 to obtain a total score ranging from 0 to 100, with higher scores indicating greater diabetes-related distress. Severe diabetes-related distress is defined as a PAID-20 total score ≥ 40. The primary endpoint is the proportion of participants with PAID-20 ≥ 40.

SECONDARY OUTCOMES:
Prevalence of severe diabetes-related distress by care setting (ambulatory vs hospitalized) | Baseline (single assessment during usual care visit, within 3 days from inclusion)
  Using the PAID-20 total score (0-100; higher scores indicate greater distress, severe distress defined as ≥ 40), the proportion of participants with severe diabetes-related distress will be calculated in two predefined subgroups: ambulatory patients (outpatient clinic and day hospital) and hospitalized patients (conventional hospitalization in endocrinology).
Factors associated with diabetes-related distress (PAID-20 score) | Baseline (single assessment during usual care visit, within 3 days from inclusion)
  The PAID-20 total score (0-100; higher scores indicate greater diabetes-related distress) will be analysed as a continuous variable. Decision-tree models (CHAID/CRT) will be used to explore associations between diabetes-related distress and predefined clinical, psychosocial and lifestyle variables.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe CAROLI-BOSC, Dr, Principal Investigator — Centre Hospitalier Universitaire de Nice

IPD SHARING:
Plan to Share IPD: Undecided